CLINICAL TRIAL: NCT02360813
Title: Randomised Controlled Trial to Evaluate the Efficacy of Cognitive Remediation Within a Secure Forensic Setting for Schizophrenia Spectrum Patients
Brief Title: Cognitive Remediation Therapy Within a Secure Forensic Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Mental Hospital (Other Government)
Responsible Party: Principal Investigator, Ken O'Reilly, Dr Ken O'Reilly. Senior Clinical Psychologist, Central Mental Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Central Mental Hospital
Record Dates: First submitted 2015-02-04; First posted 2015-02-11 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Cognitive Deficits
Keywords: Cognitive remediation therapy; Psychiatric rehabilitation; Forensic mental health; Forensic psychiatry; Clinical psychology; Randomized controlled trial; Principle driven intervention; Psychological Intervention; Cognitive enhancement
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognition Disorders | interventions — Cognitive Training; Therapeutics; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Remediation Therapy (Experimental): Principle driven cognitive remediation therapy, cognitive rehabilitation, cognitive training, cognitive enhancement.
  Interventions: Behavioral: Cognitive Remediation Therapy
- Treatment as Usual (Active Comparator): Usual care.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — Fifty-six sessions of principle driven cognitive remediation therapy. Three individual sessions and one group session each week for approximately fourteen weeks.
  Other Names: Cognitive training; Cognitive rehabilitation; Cognitive enhancement
  Arms: Cognitive Remediation Therapy
Other: Treatment as usual — Keep getting usual care.
  Other Names: Standard care
  Arms: Treatment as Usual

SUMMARY:
This clinical trial tests the feasibility, effectiveness and patient satisfaction with cognitive remediation therapy for patients diagnosed with schizophrenia or schizoaffective disorder within a forensic hospital. It is hypothesised that patients receiving cognitive remediation therapy will have an improvement in cognitive performance, real world functioning, symptoms, violence risk and benefit more from additional psychosocial treatment programmes over time relative to patients receiving treatment as usual. Furthermore it is hypothesised that it will be feasible to carry out such a study and that patients will report high rates of satisfaction with cognitive remediation therapy. Finally it is hypothesised that differences on the effectiveness measures will be maintained at 6 month follow up after the end of treatment.

DETAILED DESCRIPTION:
This is a single centre randomised clinical trial to evaluate the feasibility, effectiveness and patient satisfaction with cognitive remediation therapy within a secure forensic setting for patients diagnosed with schizophrenia or schizoaffective disorder.

The feasibility of the intervention will be assessed using key indicators such as rate of enrolment, retention of patients in the trial, blinding effectiveness, and completion rate of the primary outcome measure. The effectiveness of the intervention will be assessed using the MATRICS consensus cognitive battery, symptoms (PANSS and CAINS) and real world functioning (SOFAS: Social and occupational functioning assessment scale). The effect of cognitive remediation on violence risk (HCR-20), programme completion and recovery (Dundrum 3 & 4) will also be examined, where programme completion is a measure of attainments from participating in additional psychosocial interventions and recovery is a measure of stability of mental state.

Patient satisfaction with cognitive remediation therapy will be assessed using a consumer constructed interview developed by Rose et al (2008) and administered by a social worker not involved in the delivery of cognitive remediation.

The trial will take place at the Republic of Ireland's Central Mental Hospital (CMH). The CMH is the only secure forensic psychiatric hospital for the Republic of Ireland, a population of 4.6 million. CMH provides specialised care for adults who have a mental disorder and are at risk of harming themselves or others.

After a baseline assessment to ensure eligibility and to obtain consent, an estimated 60 patients will be randomised to receive fourteen weeks of cognitive remediation versus treatment as usual. Patients who receive treatment as usual will be offered cognitive remediation upon completion of the study. Patients allocated to cognitive remediation will receive three individual sessions of cognitive remediation a week and one group session, fifty-six sessions in total The focus of the group session is to normalise cognitive difficulties that patients may be experiencing, to receive support and to help generalise gains. The primary outcome measure the MATRICS composite score and secondary outcome measures to assess real world functioning, symptoms, violence risk, programme completion and recovery will be administered at baseline, the end of treatment and at six month follow up. Secondary measures will also include feasibility outcomes and patient satisfaction with cognitive remediation therapy. All evaluators of the effectiveness measures will be blind to participant treatment condition at the time of assessment.

The cognitive remediation therapy is a principle driven intervention consisting of nine treatment principles: Principle 1 refers to relationship building, Principle 2 refers to collaborative goal setting, Principle 3 involves the session structure, Principle 4 concerns the content of the sessions, Principle 5, concerns the pacing of sessions, Principle 6 involves scaffolding and errorless learning, Principle 7 refers to meta-cognitive strategies, Principle 8 involves generalisation of gains, finally Principle 9 refers to managing ambivalence. The actual therapy will involve the use of a combination on pen, paper and computerised materials to stimulate patient's cognitive capacity and to provide them with the opportunity to apply meta-cognitive strategies.

The investigators hypothesise that it is feasible to carry out a randomised controlled trial within a single centre forensic setting and that patients will report high rates of satisfaction with cognitive remediation. It is also hypothesised that patients receiving cognitive remediation therapy will have an improvement in cognitive performance (the primary outcome measure), real world functioning, symptoms and violence risk over time relative to patients receiving treatment as usual; specifically that there will be a treatment by time interaction. Furthermore it is hypothesised that these differences will be maintained at six month follow up after the end of treatment.

In addition it is hypothesised that patients receiving cognitive remediation will show an improvement over time on the Dundrum programme completion and recovery scales compared to those receiving treatment as usual.

While meta-analytic reviews have demonstrated that cognitive remediation therapy has a beneficial effect on the cognitive deficits experienced by patients with schizophrenia (Wykes et al 2011), to the best of our knowledge there has been no study with forensic mental health patients. The current study will help answer whether it is feasible to deliver cognitive remediation within a forensic mental health setting and whether it is acceptable to patients. The study aims to contribute to the evidence base for psychological interventions within a forensic setting and to answer the question as to whether cognitive remediation has a beneficial effect and if it does whether this effect is maintained over time.

ELIGIBILITY:
Inclusion Criteria:

* A Structured Clinical Interview for Diagnostic and Statistical Manual IV (SCID) diagnosis of schizophrenia or schizoaffective disorder.

Exclusion Criteria:

* Acutely psychotic, or judged too dangerous to participate in treatment, or being over 65 years of age.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The MATRICS Consensus Cognitive Battery (MCCB) | Group by time interaction: changes from baseline, to end of treatment (average 5 months)
  Consensus neuropsychological assessment battery for cognitive deficits in schizophrenia

SECONDARY OUTCOMES:
Social and Occupational Functioning Assessment Scale (SOFAS) | Group by time interaction: changes from baseline, to end of treatment (average 5 months)
  100 item rating scale for measuring real world functioning independent of symptoms
Positive and Negative Syndrome Scale (negative and disorganized factors) | Group by time interaction: changes from baseline, to end of treatment (average 5 months)
  Rating scale for assessing psychiatric symptoms associated with schizophrenia
Clinical Assessment Interview for Negative Symptoms (CAINS) | Group by time interaction: changes from baseline, to end of treatment (average 5 months)
  Rating scale for assessing the negative symptoms of schizophrenia

OTHER OUTCOMES:
Historical Clinical and Risk Management -20 (HCR-20) | Group by time interaction: changes from baseline, to 12 months
  Rating scale for assessing violence risk
Dundrum Toolkit: Programme Completion and Recovery Scales | Group by time interaction: changes from baseline to 12 months
  Rating scale for assessing progress and recovery within a forensic mental health setting
Patient satisfaction. | Average 5 months.
  Consumer developed interview exploring patient satisfaction with cognitive remediation.
Feasibility outcome: rate of enrolment. | 12 months.
  Willingness of forensic mental health patients to participate in study.
Feasibility outcome: rate of retention. | 12 months.
  Number of patients who complete the intervention.
Feasibility outcome: blinding. | 12 months.
  Number of patients in which the blind is broken compared to number of patients in the study.
Completion rate of primary outcome measures | 12 months.
  Number of successfully completed primary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Harry G Kennedy, M.D., Study Director — Central Mental Hospital and Department of Psychiatry, Trinity College Dublin.; Professor Gary Donohoe, Ph.D., Study Director — Department of Psychiatry, Trinity College Dublin.; Dr. Ken W O'Reilly, D.Psych.Sc., Principal Investigator — Central Mental Hospital and Department of Psychiatry, Trinity College Dublin.
Locations (1):
- Central Mental Hospital, Dublin, Ireland

REFERENCES:
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Rybarczyk B. (2011). Social and Occupational Functioning Assessment Scale (SOFAS). Encyclopedia of Clinical Neuropsychology. p 2313
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Kring AM, Gur RE, Blanchard JJ, Horan WP, Reise SP. The Clinical Assessment Interview for Negative Symptoms (CAINS): final development and validation. Am J Psychiatry. 2013 Feb;170(2):165-72. doi: 10.1176/appi.ajp.2012.12010109. PMID 23377637
- [Background] Webster CD, Douglas KS, Eaves D, Hart SD. HCR-20: assessing risk for violence. Burnaby: Mental Health Law and Policy Institute, Simon Fraser University; 1997.
- [Background] Davoren M, Abidin Z, Naughton L, Gibbons O, Nulty A, Wright B, Kennedy HG. Prospective study of factors influencing conditional discharge from a forensic hospital: the DUNDRUM-3 programme completion and DUNDRUM-4 recovery structured professional judgement instruments and risk. BMC Psychiatry. 2013 Jul 9;13:185. doi: 10.1186/1471-244X-13-185. PMID 23837697
- [Background] Rose D, Wykes T, Farrier D, Doran AM, Sporel T & Bogner D (2008) What Do Clients Think of Cognitive Remediation Therapy?: A Consumer-Led Investigation of Satisfaction and Side Effects, American Journal of Psychiatric Rehabilitation. Rehabilitation, 11:2, 181-204.
- [Background] Wykes T, Huddy V, Cellard C, McGurk SR, Czobor P. A meta-analysis of cognitive remediation for schizophrenia: methodology and effect sizes. Am J Psychiatry. 2011 May;168(5):472-85. doi: 10.1176/appi.ajp.2010.10060855. Epub 2011 Mar 15. PMID 21406461
- [Derived] O'Reilly K, Donohoe G, O'Sullivan D, Coyle C, Corvin A, O'Flynn P, O'Donnell M, Galligan T, O'Connell P, Kennedy HG. A randomized controlled trial of cognitive remediation for a national cohort of forensic patients with schizophrenia or schizoaffective disorder. BMC Psychiatry. 2019 Jan 15;19(1):27. doi: 10.1186/s12888-019-2018-6. PMID 30646884
- [Derived] O'Reilly K, Donohoe G, O'Sullivan D, Coyle C, Mullaney R, O'Connell P, Maddock C, Nulty A, O'Flynn P, O'Connell C, Kennedy HG. Study protocol: a randomised controlled trial of cognitive remediation for a national cohort of forensic mental health patients with schizophrenia or schizoaffective disorder. BMC Psychiatry. 2016 Jan 13;16:5. doi: 10.1186/s12888-016-0707-y. PMID 26759167